CLINICAL TRIAL: NCT07284290
Title: Elucidating the Role of Cholinergic Degeneration in Cognitive Fluctuations in Lewy Body Dementia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HM20033370; R01NS142622 (NIH)
Record Dates: First submitted 2025-12-10; First posted 2025-12-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Dementia With Lewy Bodies; Parkinson Disease Dementia; Healthy Controls
Keywords: Parkinson Disease with Mild Cognitive Impairment; Mild Cognitive Impairment with Lewy Bodies
MeSH Terms: conditions — Lewy Body Disease

STUDY DESIGN:
Intervention Model Description: A cross-sectional case control study in which cholinergic degeneration in 45 subjects with DLB or PDD with CF will be compared to a group of 45 subjects with Lewy Body disease without CF and 30 healthy controls. The first 20 participants who are eligible and consent will also participate in an 8-week pre-post interventional cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Subjects with DLB or PDD (Experimental): 90 subjects with Dementia with Lewy Bodies (DLB) or Parkinson's Disease with Dementia (PDD)
  Interventions: Procedure: Syn-One skin biopsy; Diagnostic Test: Multi modal MRI; Diagnostic Test: Assessment of dynamic EEG features over 48-hour periods across all study aims; Diagnostic Test: Plasma biomarkers
- Subjects with Lewy Body disease with CF (Active Comparator): A subset of 20 subjects with Lewy Body (LB) disease with Cognitive fluctuations (CF)
  This arm will be a subset of 20 subjects from Arm #1 (Subjects with DLB or PDD).
  Interventions: Diagnostic Test: Multi modal MRI; Diagnostic Test: Assessment of dynamic EEG features over 48-hour periods across all study aims; Drug: Galantamine HBr extended-release 8mg capsules (8mg ER).
- Healthy control subjects (Other): 30 healthy controls
  Interventions: Diagnostic Test: Multi modal MRI; Diagnostic Test: Assessment of dynamic EEG features over 48-hour periods across all study aims; Diagnostic Test: Plasma biomarkers

INTERVENTIONS:
Procedure: Syn-One skin biopsy — Detects phosphorylated alpha synuclein in cutaneous nerve fibrils which has >95% sensitivity in detecting DLB
  Arms: Subjects with DLB or PDD
Diagnostic Test: Multi modal MRI — Functional MRI used to investigate the network connectivity changes associated with alterations in the cholinergic system. Using this comprehensive methodology to establish cholinergic degeneration's contribution to CF provides a robust framework for future research and therapeutic strategies.
Diagnostic Test: Assessment of dynamic EEG features over 48-hour periods across all study aims — Implementing prolonged EEG monitoring, to capture dynamic changes in neural activity associated with CF. The methods are designed avoid the limitations identified in a systematic review of EEG studies in DLB, as will use quantitative analysis of EEG, uniformly apply diagnostic criteria, and consider the confounding effects of medications.
  Concurrent evaluation of PVT performance and EEG This dual assessment will correlate cognitive and neurophysiological dynamics in real-time, providing a more holistic understanding of CF over time and the functional brain activity that underlies them. Temporal integration of PVT with EEG data collection will enable the identity of specific correlates of CF.
Diagnostic Test: Plasma biomarkers — A blood sample will be collected and sent for processing by C2N Diagnostics for the detection of Aβ42/40 and p-tau217 via mass spectrometry, a method shown to be highly accurate for predicting amyloid positivity on PET (AUC=0.94). Exploratory Biomarkers: The additional blood sample will be used for analysis of exploratory biomarkers and future research. A total of up to 20mL of blood will be taken.
  Arms: Healthy control subjects; Subjects with DLB or PDD
Drug: Galantamine HBr extended-release 8mg capsules (8mg ER). — 20 participants from the arm 1. Participants will take 1 capsule daily of galantamine 8mg ER for 4 weeks and then increase to 2 capsules daily of galantamine 8mg ER (16mg) for 4 weeks. This titration will mitigate potential for cholinergic side effects. At 2 weeks, 4 weeks and 6 weeks of the treatment period, safety and compliance will be assessed during phone call visits. Any adverse event rated as Grade 2 or greater according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 and that is definitely or possibly attributable to the study drug will result in study drug withdrawal or dose reduction.
  Arms: Subjects with Lewy Body disease with CF

SUMMARY:
The proposed study aims to address the critical gaps in understanding the mechanisms of CF (Cognitive Fluctuations) by leveraging recently emerged molecular biomarkers, advanced neuroimaging techniques to assess measures of cholinergic degeneration, and synchronous EEG and assessments of attention. One of the overarching innovations of study is combining all of these assessments into one integrated research plan

DETAILED DESCRIPTION:
Aim 1 is a cross-sectional case control study in which cholinergic degeneration in 45 participants with DLB or PDD with CF will be compared to a group of 45 individuals with Lewy Body disease without CF and 30 healthy controls. The first 20 participants who are eligible for Aim 2 and consent will also participate in an 8-week pre-post interventional cohort study immediately following Aim 1 procedures. For Aim 3, Aim 1 participants will complete annual follow-up evaluations for 2 years to understand factors influencing the change in cognitive fluctuations over time.

ELIGIBILITY:
Inclusion Criteria:

Arm 1:

* Age range: 50 ≤ age < 90.
* Diagnosis of dementia with Lewy bodies (DLB), Parkinson disease dementia (PDD), Parkinson disease with Mild Cognitive Impairment (PD-MCI), Mild Cognitive Impairment with Lewy bodies (MCI-LB).
* DLB participants must fulfill criteria for clinically probable DLB based on the 2017 4th consensus report of the DLB consortium.
* PDD participants must meet criteria for clinically probable PD according to the MDS Clinical Diagnostic Criteria for Parkinson's Disease and must also meet criteria for probable PDD based on the 2007 Movement Disorders Society clinical diagnostic criteria.
* PD-MCI participants must meet criteria for clinically probable PD according to the MDS Clinical Diagnostic Criteria for Parkinson's Disease and meet criteria for Mild Cognitive Impairment on cognitive testing at screening.
* MCI-LB participants with must meet established research criteria.
* Capacity to provide informed consent or, if unable, availability of a legally authorized representative or guardian who can provide informed consent.
* Availability of informant (for participants meeting criteria for dementia).
* Ability and willingness to comply with the study-related procedures.
* Fluent in spoken and written English (due to cognitive testing)

Exclusion Criteria:

Arm 1

* History of cognitive disorder or psychiatric disorder other than that related to dementia with Lewy bodies or Parkinson disease dementia.
* History of deep brain stimulation or any neurosurgical procedure.
* History of structural brain disease or known significant cerebrovascular disease.
* History of seizures or epilepsy and/or use of sodium channel blockers, i.e. carbamazepine, oxcarbazepine, phenytoin, topiramate, lamotrigine, felbamate, zonisamide, rufinamide, lacosamide, eslicarbazepine, and valproate.
* Greater than two alcoholic drinks per day for men and one per day for women.
* Regular use of benzodiazepines or barbiturates. (If benzodiazepines are taken as needed only, these medications cannot be taken within 5 half-lives of screening visit or between screening visit and EEG.)
* Severe dementia (based on PI assessment of subject dependence level for instrumental activities of daily living)
* Any contraindication to brain MRI.
* Any medical condition that would interfere with ability to complete all study procedures.
* Participants must not be pregnant, planning to become pregnant, or father a child for the duration of the study

Inclusion Criteria:

Arm 2 (Cholinesterase inhibitor cohort) inclusion criteria:

* Completed Aim 1.
* Clinical diagnosis of LBD (DLB or PDD) with CF.
* Not taking a cholinesterase inhibitor and has not taken a cholinesterase inhibitor in the previous 90 days.
* Ability and willingness to comply with the ChEI Cohort procedures (including galantamine administration), or a caregiver willing and able to ensure compliance.

Exclusion Criteria:

Arm 2 (Cholinesterase inhibitor cohort) exclusion criteria:

* Severe hepatic impairment.
* Renal failure.
* Significant bradycardia (<50 bpm) at screening or history of AV block.
* Any contraindication to galantamine administration based on PI discretion.

Inclusion criteria:

Arm 3 (Healthy Controls)

* Age range: 50 ≤ age < 90.
* Healthy controls should not have any known neurologic conditions that could interfere with study procedures or results.
* Capacity to provide informed consent or, if unable, availability of a legally authorized representative or guardian who can provide informed consent.
* Availability of informant (for participants meeting criteria for dementia).
* Ability and willingness to comply with the study-related procedures.
* Fluent in spoken and written English (due to cognitive testing).

Exclusion Criteria:

Arm 3 (Healthy Controls)

* No History of cognitive disorder or psychiatric disorder other than that related to dementia with Lewy bodies or Parkinson disease dementia.
* No History of deep brain stimulation or any neurosurgical procedure.
* No History of structural brain disease or known significant cerebrovascular disease.
* No History of seizures or epilepsy and/or use of sodium channel blockers, i.e. carbamazepine, oxcarbazepine, phenytoin, topiramate, lamotrigine, felbamate, zonisamide, rufinamide, lacosamide, eslicarbazepine, and valproate.
* Any medical condition that would interfere with ability to complete all study procedures.
* Participants must not be pregnant, planning to become pregnant, or father a child for the duration of the study

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Clinical Assessment of Fluctuations (CAF) (frequency and duration score) | Screening, Baseline, ChEI Cohort Day 56, 1 year follow-up visit, and 2 year follow-up visit
  The scoring for the Clinical Assessment of Fluctuations (CAF) is a two-step process that uses both a frequency and a duration score. The two scores are multiplied together to get the final severity rating. A higher score indicates more severe cognitive fluctuations. After rating the frequency and duration, the two scores are multiplied to get the final CAF score.
  Frequency score x Duration score=Total CAF score
Dementia Cognitive Fluctuations Scale-Research Version (DCFS-R) (total score) | Screening, Baseline, ChEI Cohort Day 56, 1 year follow-up visit, and 2 year follow-up visit
  The DCFS-R is measured as a total score from 4 to 20, with higher scores indicating more severe cognitive fluctuations in dementia. It is calculated by summing a nurse's ratings on four items, each scored on a 5-point Likert scale (1=no difference, 5=very large difference). The four items assess the difference between a person's best and worst functioning, which includes daytime somnolence, drowsiness, and altered levels of consciousness.
Mayo Fluctuations Scale (Four questions) | Screening, Baseline, ChEI Cohort Day 56, 1 year follow-up visit, and 2 year follow-up visit
  The four questions included in the Mayo Fluctuations Scale have been found to significantly differentiate Alzheimer's Disease from DLB. Positive items are summed to create a "fluctuations composite score" with a score of 3 or 4 associated with DLB.
Functional Activities Questionnaire (FAQ Assessment) | Screening, Baseline, 1 year follow-up visit, and 2 year follow-up visit
  The FAQ is a number from 0 to 30 that represents a person's independence in daily tasks, with higher scores indicating more difficulty. The score is calculated by summing the ratings (0-3) for 10 activities, and a cut-off score of 9 or higher is often used to suggest potential cognitive or functional impairment.
Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) | Screening, Baseline, 1 year follow-up visit, and 2 year follow-up visit
  The MDS-UPDRS is a tool that measures the experiences of daily living (Part I), motor experiences of daily living (Part II), motor examination (Part III), and motor complications (Part IV). Scores range from 0 to 260, with 0 indicating no disability and higher scores indicating greater disability. The individual parts are rated on a scale of 0 to 4, with higher scores indicating greater impairment.
REM Sleep Behavior Disorder Questionnaire (RBDSQ) | Screening, Baseline, 1 year follow-up visit, and 2 year follow-up visit
  The RBDSQ is measured by a total from 0-13, with a score of 5 or higher indicating a positive result for REM Sleep Behavior Disorder (RBD). The questionnaire is a 10-item self-rating tool to screen for RBD, and the cutoff score can vary depending on the population being screened.
Neuropsychiatric Inventory (NPI) | Screening, Baseline, 1 year follow-up visit, and 2 year follow-up visit
  The NPI is an interview performed with a caregiver to assess any changes in the participants' behavior related to delusions, hallucinations, anxiety, and apathy. It is comprised of 4 main questions, 31 sub-questions and frequency/severity ratings.
Enhanced Scale for the assessment for Parkinson's Disease (SAPS-PD) | Screening, Baseline, 1 year follow-up visit, and 2 year follow-up visit
  The eSAPS-PD is used to measure the severity of hallucinations and delusions in patients with Parkinson's Disease Psychosis (PDP). Scored on a scale of 0 to 5 for each of its 9 items, resulting in a total score from 0 to 45. Each item is rated based on the severity of the symptom, with a score of 0 meaning "None" and a score of 5 meaning "Severe".
Patient Health Questionnaire-9 (PHQ-9) | Screening, Baseline, 1 year follow-up visit, and 2 year follow-up visit
  The PHQ-9 is a self-report measure used to screen for and assess the severity of depression in adults. It consists of nine questions based on the diagnostic criteria for major depressive disorder in the DSM-5. The total score for the PHQ-9 can range from 0 to 27. Each of the nine items is scored based on the frequency with which a person has experienced a specific symptom over the past two weeks: 0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day. The scores for all nine items are added together to produce a total severity score. While scores of 10 or higher have high sensitivity and specificity for identifying major depression, the PHQ-9 alone is not a diagnostic tool. A clinical interview is necessary for a definitive diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Barrett, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No